CLINICAL TRIAL: NCT00557466
Title: A Randomized, Multi-center, Parallel Group, Double Blind, Placebo and Formoterol Controlled 14 Day Dose Ranging Trial of 4 Doses of Indacaterol Delivered Via TWISTHALER® Device in Patients With COPD
Brief Title: A Dose Ranging Trial of 4 Doses of Indacaterol Delivered Via the TWISTHALER® Device in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149B2201
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: QMF; indacaterol; TWISTHALER® device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- indacaterol 62.5 μg (Experimental): Indacaterol 62.5 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2- agonist
- indacaterol 125 μg (Experimental): Indacaterol 125 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2- agonist
- Indacaterol 250 μg (Experimental): Indacaterol 250 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2- agonist
- indacaterol 500 μg (Experimental): Indacaterol 500 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: indacaterol; Drug: placebo to formoterol; Drug: short acting β2- agonist
- formoterol (Active Comparator): Formoterol 12 μg delivered by the AEROLIZER® device twice a day and placebo to indacaterol (placebo TWISTHALER® device) once a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: formoterol; Drug: placebo to indacaterol; Drug: short acting β2- agonist
- placebo (Placebo Comparator): Placebo to indacaterol (placebo TWISTHALER® device) once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days. All participants were supplied with salbutamol/albuterol to use throughout the study as rescue medication.
  Interventions: Drug: placebo to indacaterol; Drug: placebo to formoterol; Drug: short acting β2- agonist

INTERVENTIONS:
Drug: indacaterol — Indacaterol delivered by multiple dose dry powder inhaler (TWISTHALER® device).
  Arms: Indacaterol 250 μg; indacaterol 125 μg; indacaterol 500 μg; indacaterol 62.5 μg
Drug: formoterol — Formoterol delivered by oral inhalation via AEROLIZER® inhalation device.
  Arms: formoterol
Drug: placebo to indacaterol — Placebo TWISTHALER® device
  Arms: formoterol; placebo
Drug: placebo to formoterol — Placebo AEROLIZER® device
  Arms: Indacaterol 250 μg; indacaterol 125 μg; indacaterol 500 μg; indacaterol 62.5 μg; placebo
Drug: short acting β2- agonist — 100 μg / 90 μg salbutamol/albuterol Metered Dose Inhaler (MDI) or equivalent dose of Dry Powder Inhaler (DPI).

SUMMARY:
This study will evaluate the dose response relationship among four doses of indacaterol as well as placebo delivered via the TWISTHALER® device.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure (which include any adjustment to their current COPD treatment)
* Cooperative outpatients with a diagnosis of COPD (moderate to severe as classified by the Global Initiative for Obstructive Lung Disease (GOLD) Guidelines, 2006) and:

  * Smoking history of at least 10 pack years
  * Post-bronchodilator Forced Expiratory Volume in one second (FEV1) < 80% and ≥30% of the predicted normal value.
  * Post-bronchodilator FEV1/Forced vital capacity (FVC) < 70%

Exclusion Criteria:

* Pregnant women, nursing mothers, or females of childbearing potential, regardless of whether or not sexually active, if they are not using acceptable methods of contraception.
* Patients who have been hospitalized for an exacerbation of their airways disease within 6 weeks prior to Visit 1 or between Visit 1 and Visit 2.
* Patients with a history of asthma.
* Patients with an acute respiratory tract infection within 4 weeks prior to Visit 1, will be not allowed to enter the study.
* Other clinically significant conditions which may interfere with the study conduct or patient safety as specified in the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (75):
- Argentina (3):
  - Novartis Investigator site, Buenos Aires
  - Novartis Investigator Site, Rosario
  - Novartis Investigator Site, Santillán
- Novartis Investigator Site, Liège, Belgium
- Chile (2):
  - Novartis Investigator Site, Santiago
  - Novartis Investigator Site, Val Pariso
- France (6):
  - Novartis Investigator Site, Bois-Guillaume
  - Novartis Investigator Site, Clermot Ferand
  - Novartis Investigator Site, Lille
  - Novartis Investigator Site, Marseille
  - Novartis Investigator Site, Nantes
  - Novartis Investigator site, Toulouse
- Germany (11):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator site, Bibertal
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site - 2 sites, Bonn
  - Novartis Investigator Site, Cologne
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Heidelberg
  - novartis Investigator site, Koblenz
  - Novartis Investigator Site, Marburg
  - Novartis Investigator Site, Solingen
- Hungary (3):
  - Novartis Investigator Site, Budapest
  - Novartis Investigator Site, Debrecen
  - Novartis investigator site, Pécs
- Novartis investigator site, Dublin, Ireland
- Italy (3):
  - Novartis Investigator Site, Genova
  - Novartis Investigator Site, Napoli
  - Novartis Investigator Site, Pordenone
- Latvia (2):
  - Novartis investigator site, Daugavpils
  - Novartis Investigator Site, Riga
- Lithuania (3):
  - Novartis Investigator Site, Kaunas
  - Novartis Investigator Site, Klaipėda
  - Novartis Investigator Site, Vilnius
- Novartis Investigator Site, Tronheim, Norway
- Novartis Investigator Site, Lima, Peru
- Poland (8):
  - Novartis Investigator Site, Izabelin
  - Novartis Investigator Site, Lodz
  - Novartis Investigator Site, Lublin
  - Novartis Investigator site, Mrozy
  - Novartis Investigator Site, Olsztyn
  - Novartis Investigator Site, Rzeszów
  - Novartis Investigator Site, Wejhrowo
  - Novartis Investigator Site, Włocławek
- Romania (4):
  - Novartis Investigator Site, Bucharest
  - Novartis Investigator Site, Cluj-Napoca
  - Novartis Investigator Site, Iași
  - Novartis Investigator Site, Timișoara
- South Africa (10):
  - Novartis Investigator Site, Bloemfontain
  - Novartis Investigator Site, Bloemfontein
  - Novartis Investigator Site, Cape Town
  - Novartis Investigator Site, Durban
  - Novartis Investigator Site, eManzimtoti
  - Novartis Investigator Site, George
  - Novartis Investigator Site, Johannesburg
  - Novartis Investigator Site, Port Elizabeth
  - Novartis Investigator Site, Pretoria
  - Novartis Investigator Site, Tygerberg
- Turkey (Türkiye) (9):
  - Novartis Investigator Site, Erzurum
  - Novartis Investigator Site, Isparta
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Kahramanmaraş
  - Novartis Investigator Site, Kayseri
  - Novartis Investigator Site, Malatya
  - Novartis Investigator Site, Manisa
  - Novartis Investigator Site, Sanliurfa
  - Novartis Investigator Site, Trabzon
- United Kingdom (7):
  - Novartis Investigator Site, Belfast
  - Novartis Investigator Site, Chesterfield
  - Novartis Investigator Site, Glasgow
  - Novartis Investigator Site, Plymouth
  - Novartis Investigator Site, Warminster
  - Novartis investigator site, Watford
  - Novartis Investigator Site, Whitstable

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol 62.5 μg: Indacaterol 62.5 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 125 μg: Indacaterol 125 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 250 μg: Indacaterol 250 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Indacaterol 500 μg: Indacaterol 500 μg delivered by the TWISTHALER® device once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
- Formoterol: Formoterol 12 μg delivered by the AEROLIZER® device twice a day and placebo to indacaterol (placebo TWISTHALER® device) once a day for 14 days.
- Placebo: Placebo to indacaterol (placebo TWISTHALER® placebo) once a day and placebo to formoterol (placebo AEROLIZER® device) twice a day for 14 days.
Period: Overall Study
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Started | 98 | 92 | 101 | 96 | 90 | 91
Safety Population | 98 (All randomized patients who received at least one dose of the study drug) | 92 (All randomized patients who received at least one dose of the study drug) | 101 (All randomized patients who received at least one dose of the study drug) | 96 (All randomized patients who received at least one dose of the study drug) | 90 (All randomized patients who received at least one dose of the study drug) | 91 (All randomized patients who received at least one dose of the study drug)
Intent to Treat Population | 98 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement) | 91 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement) | 98 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement) | 93 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement) | 87 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement) | 89 (All randomized patients who had a baseline and at least one post-dose FEV1 measurement)
Completed | 94 | 87 | 95 | 92 | 87 | 85
Not Completed | 4 | 5 | 6 | 4 | 3 | 6
Not completed — Adverse Event | 3 | 1 | 4 | 1 | 2 | 4
Not completed — Abnormal laboratory value(s) | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Subject withdrew consent | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Administrative problems | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Abnormal test procedure results | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo | Total
Number analyzed (Participants) | 98 | 91 | 98 | 93 | 87 | 89 | 556
Age Continuous [Mean (Standard Deviation); unit: years] — Total number of baseline participants is based on the Intent to Treat Population
  years | 62.1 (7.69) | 61.6 (9.51) | 61.6 (8.68) | 61.9 (8.48) | 63.3 (8.36) | 62.2 (8.84) | 62.1 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 23 | 27 | 20 | 29 | 25 | 157
  Male | 65 | 68 | 71 | 73 | 58 | 64 | 399

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from baseline to 24 hour post dose trough FEV1 after 14 days of treatment was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Baseline (prior to first dose) and Day 15 (24 hours after last dose)
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. The analysis only includes patients with non-missing data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 92 | 85 | 90 | 89 | 83 | 80
liters | 0.051 (0.0207) | 0.073 (0.0217) | 0.076 (0.0210) | 0.121 (0.0211) | 0.098 (0.0219) | 0.005 (0.0223)

2. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) Between Baseline (Predose) and 4 Hours Post-dose
Description: FEV1 was measured on Day 14 pre-dose and up to 4 hours post-dose. The Area Under the Curve (AUC) for FEV1 was analyzed using Analysis of Covariance adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 14, pre-dose and at 5, 20, 30 minutes and 1, 2, 3, and 4 hours post-dose.
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. Observed data only.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 93 | 86 | 90 | 89 | 83 | 81
liters | 1.407 (0.0193) | 1.461 (0.0202) | 1.441 (0.0196) | 1.500 (0.0198) | 1.541 (0.0206) | 1.315 (0.0208)

3. Secondary Outcome: The Mean Change From Baseline to 24 Hour Post-dose (Trough) Forced Expiratory Volume in 1 Second (FEV1) on Day 1
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Change from baseline to 24 hour post dose trough FEV1 after 1 day of treatment was analyzed using Analysis of Covariance (ANCOVA) adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 1 Baseline (prior to first dose) and 24 hours post-dose.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 95 | 88 | 96 | 90 | 86 | 87
liters | 0.028 (0.0152) | 0.054 (0.0158) | 0.060 (0.0151) | 0.073 (0.0156) | 0.140 (0.0160) | -0.009 (0.0160)

4. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) Between Baseline (Predose) and 4 Hours Post-dose on Day 1
Description: FEV1 was measured on Day 1 pre-dose and up to 4 hours post-dose. The Area Under the Curve (AUC) for FEV1 was analyzed using Analysis of Covariance adjusting for treatment and region with baseline FEV1 as a covariate.
Time Frame: Day 1; pre-dose and at 5, 20, 30 minutes and 1, 2, 3, and 4 hours post-dose.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 98 | 91 | 97 | 91 | 87 | 87
liters | 1.371 (0.0111) | 1.422 (0.0116) | 1.427 (0.0112) | 1.438 (0.0116) | 1.535 (0.0118) | 1.321 (0.0118)

5. Secondary Outcome: Time to Peak Forced Expiratory Volume in 1 Second (FEV1) on Day 1 and Day 14
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Time to peak FEV1 is calculated in minutes from the time of inhalation of study drug to the time of the peak FEV1, which is taken as the maximum FEV1 recorded post-dose.
Time Frame: Day 1 and Day 14 measured pre-dose and up to 4 hours post-dose
Population: The intent-to-treat population (ITT) population consisted of all randomized patients who had a baseline and at least one post-dose FEV1 measurement. The analysis only includes patients with non-missing data, indicated by "N".
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 98 | 91 | 98 | 93 | 87 | 89
minutes
  Day 1 [N=98, 91, 97, 91, 87, 87] | 80.9 (76.01) | 84.4 (77.74) | 101.4 (83.44) | 105.3 (81.85) | 115.0 (81.59) | 85.7 (81.44)
  Day 14 [N=93, 86, 90, 89, 83, 82] | 91.3 (81.20) | 105.6 (82.53) | 104.7 (75.96) | 116.4 (85.03) | 89.1 (72.91) | 68.0 (70.38)

6. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow
Description: The Peak Expiratory Flow (PEF) rate is the maximal rate that a person can exhale during a short maximal expiratory effort after fully inhaling. Participants measured their PEF using a peak flow meter prior to taking study medication and recorded measurements in a diary every morning and evening during the study. Change from baseline is the difference between the mean baseline PEF recorded during the screening period until the first day of treatment, and the overall mean PEF from Days 1 to 14.
Time Frame: Baseline (recorded during the screening period) and Days 1-14 (treatment period).
Population: Intent to treat population. The analysis only includes patients with non-missing data.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 98 | 91 | 98 | 93 | 87 | 89
liters/minute
  Morning [N=56, 63, 59, 54, 54, 55] | 3.10 (29.709) | 19.91 (34.060) | 23.63 (30.707) | 11.11 (36.787) | 16.06 (31.544) | -4.24 (31.357)
  Evening [N=56, 58, 56, 49, 48, 52] | -2.72 (28.816) | 13.42 (30.500) | 19.00 (24.004) | 5.92 (43.490) | 14.97 (40.355) | -2.75 (35.034)

7. Secondary Outcome: Number of Participants Using Rescue Medication
Description: Participants recorded the use of rescue medications (salbutamol/albuterol) for treatment of asthma symptoms twice a day in a diary during the 14 days of the treatment period.
Time Frame: Over 14 days
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Number analyzed (Participants) | 98 | 91 | 98 | 93 | 87 | 89
participants
  Day | 74 | 61 | 73 | 65 | 65 | 70
  Night | 72 | 60 | 67 | 59 | 67 | 72

ADVERSE EVENTS:
Arm/Group | Indacaterol 62.5 μg | Indacaterol 125 μg | Indacaterol 250 μg | Indacaterol 500 μg | Formoterol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/92 | 1/101 | 2/96 | 1/90 | 1/91
Other Adverse Events (participants affected / at risk) | 4/98 | 5/92 | 3/101 | 4/96 | 6/90 | 8/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 62.5 μg (N=98) | Indacaterol 125 μg (N=92) | Indacaterol 250 μg (N=101) | Indacaterol 500 μg (N=96) | Formoterol (N=90) | Placebo (N=91)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 62.5 μg (N=98) | Indacaterol 125 μg (N=92) | Indacaterol 250 μg (N=101) | Indacaterol 500 μg (N=96) | Formoterol (N=90) | Placebo (N=91)
NASOPHARYNGITIS (Infections and infestations) | 2 | 0 | 1 | 1 | 5 | 2
HEADACHE (Nervous system disorders) | 2 | 5 | 2 | 3 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.